CLINICAL TRIAL: NCT04890132
Title: Vestibular Precision: Physiology & Pathophysiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Richard Lewis, Associate Professor, Otolaryngology and Neurology; Director, Jenks Vestibular Laboratory, Massachusetts Eye and Ear Infirmary., Massachusetts Eye and Ear Infirmary
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019A015798
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Vestibular Schwannoma; Inner Ear Disease; Dizziness; Neurofibromatosis 2; Vestibular Disorder
Keywords: VOR variability; Vestibular Precision; Neural Noise; Motion Perception; Perceptual Precision; Vestibular Ocular Reflex
MeSH Terms: conditions — Neuroma, Acoustic; Labyrinth Diseases; Dizziness; Neurofibromatosis 2; Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Controls (Experimental): normal control participants - no history of neurologic or inner ear disease
  Interventions: Behavioral: VOR precision training
- Peripheral Vestibular Dysfunction (Experimental): Patients with unilateral vestibular damage due to monophasic illness such as vestibular neuritis or vestibular schwannoma (VS).
  For VS patients, the investigators will test them in three states: pre-op, sub-acute post-op (6 weeks), and chronic post-op (6 months).
  Interventions: Behavioral: VOR precision training

INTERVENTIONS:
Behavioral: VOR precision training — Subjects are rotated in yaw using a pseudo-random sum of sines motion (0.5 - 2.0 Hz), view a monitor 1 m away, and are instructed to move their avatar through a maze using a joystick. The size of the maze becomes smaller in real-time when they are successful so that the patient is at the limit of their acuity. This task requires patients to optimize dynamic visual acuity to threshold-level images while rotating. We predict that VOR precision will gradually improve during training and that after training VOR precision will be better than the pre-training data. The sham task is as above but the acuity required to see the maze will set at a much larger level so baseline visual precision will be adequate to perform the task easily.

SUMMARY:
This project will investigate the role of noise in the vestibular system, and in particular its effects on the variability (precision) of vestibular-mediated behaviors. The investigators will study vestibular precision in normal subjects and patients with peripheral vestibular damage, and will investigate its potential plasticity. The goals are to develop a better understanding of the role noise plays in the vestibular system in normal and pathologic populations, and to determine if the brain can learn to improve signal recognition within its inherently noisy neural environment, which would result in improved behavioral precision.

DETAILED DESCRIPTION:
The goal of this study is to investigate vestibular precision by quantifying the variability in behavioral responses that result from the neural noise inherent to the peripheral and central vestibular systems. Because neural noise contaminates the signals that are transduced by the ear and processed by the brain, vestibular-mediated behavioral responses vary even when identical stimuli are provided. In this study, the investigators focus on vestibular precision in human subjects and investigate its sources, its effects on behavior, and its degradation when the periphery is damaged and its potential plasticity. Specifically, the investigators will investigate: (1) Vestibular precision in normal subjects - physiology: A) The investigators will measure the angular and linear vestibulo-ocular reflex (VOR) using novel motion combinations that reinforce or cancel eye movement responses, which will allow us to determine the distribution and magnitude of noise produced in the sensory (canal, otolith) pathways and in the oculomotor pathway. The investigators hypothesize that normal subjects will demonstrate a bimodal distribution of noise with either sensory or motor predominance, and that subjects with more sensory noise will demonstrate other behavioral characteristics that reflect this characteristic (e.g., higher perceptual thresholds); and B) The investigators will assay vestibular noise from trial-trial variations in the VOR and will compare VOR dynamics with those predicted by a Bayesian model using the assayed noise. The investigators predict variations in VOR dynamics across subjects, age and stimulus amplitudes will be consistent with Bayesian processing of noise. Potential confounding factors will be carefully controlled, including attention, fatigue, and non-vestibular cues. (2) Vestibular precision after peripheral damage - pathophysiology: A) The investigators will examine the changes in vestibular precision that occur when one vestibular nerve is damaged (by a vestibular schwannoma, VS) and after the damaged nerve is surgically sectioned, and will investigate if precision measurements can provide evidence of pathologic noise produced by the damaged nerve and therefore help predict clinical outcome when the nerve is sectioned. The investigators hypothesize that changes in signal reliability due to the VS will be traceable to both the reduced redundancy caused by loss of afferent fibers and to aberrant noise generated by the damaged vestibular nerve and that changes in precision after neurectomy will correlate the outcome measures that characterize patient disability; and B) The investigators will examine the plasticity of vestibular precision in the oculomotor and perceptual realms with the goal of determining if precision can be improved. Using novel training approaches that provide challenging signal extraction tasks, the investigators hypothesize that participants will improve their vestibular precision on the trained task. As secondary outcome measures, the investigators will determine if training one behavior generalizes to the non-trained behavior and if patient's symptoms are affected by improved precision.

ELIGIBILITY:
Inclusion Criteria:

Normal subjects:

* normal vestibular-oculomotor exams
* normal low-frequency standard rotational testing
* normal hearing

Vestibular Schwannoma:

* existence of unilateral vestibular schwannoma (pre & post surgical resection)
* must have sub-occipital surgical approach with complete sectioning of the vestibular nerve
* rotational testing to assess pre-surgical vestibular function
* audiogram
* brain MRI consistent with vestibular schwannoma
* audiography in each ear

Exclusion Criteria:

Normal subjects

* history of otologic or neurologic disease
* on vestibular suppressant medication (benzodiazepine, antihistamine, anticholinergic)

Vestibular Schwannoma

* other otologic disease (other than presbycusis) or any neurologic disease (other than migraine)
* on vestibular suppressant medication (benzodiazepine, antihistamine, anticholinergic)

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in perceptual thresholds | baseline and post-training (1 hour)
  Measurements of motion perception thresholds (yaw for rotational tasks, roll tilt for tilt task) before and after training.
Change in rapid measure of gait | baseline and post-training (1 hour)
  This measure is scored before and after VOR precision training in UVD (unilateral vestibular dysfunction) patients. Gait is scored by performance on a task derived from the FGA (walking 40 feet while turning the head from side to side). It is scored on a 0 to 10 visual scale and provides a rapid assessment of vestibular function pre and post adaptation.
Change in measure of inducible dizziness | baseline and post-training (1 hour)
  Looking at the change between before and after VOR precision training in UVD (unilateral vestibular dysfunction) patients. Inducible dizziness is the symptom severity provoked by a task derived from the FGA (walking 40 feet while turning the head from side to side). It is scored on a 0 to 10 visual scale and provides a rapid assessment of vestibular function pre and post adaptation.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States